CLINICAL TRIAL: NCT05277714
Title: Neurofeedback Based on Near-infrared Spectroscopy as a Therapy for Food Addiction in Obese Subjects.
Acronym: CaDOb
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 35RC21_8946_08_CadOb
Record Dates: First submitted 2022-03-02; First posted 2022-03-14 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Craving
MeSH Terms: conditions — Obesity | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Masking Description: sham procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NF (Experimental)
  Interventions: Other: NF
- Sham (Sham Comparator)
  Interventions: Other: Sham

INTERVENTIONS:
Other: Sham — The sham protocol will last 15 minutes per session, and during each session, the participants will receive the same instruction but will be shown a random signal, the goal being that the control strategy that the participant tries to implement is not correlated with the visual feedback provided by the gauge.
  Arms: Sham
Other: NF — The neurofeedback protocol will be the same during the 8 sessions constituting the protocol and taking place over a period of 4 weeks (2 neurofeedback sessions per week, the first and the last one in an MRI context). It will last 15 minutes per session, and during each session, the patient will have to increase the brain activity of her dlPFC using a visual gauge representing the "activity level" of her own dlPFC. No specific instructions will be given to the volunteer so that he/she can develop his/her own internal strategy to increase this "activity level".
  Arms: NF

SUMMARY:
The hypothesis is that the increase in dlPFC brain activity via near-infrared spectroscopy-based Neurofeedback (fNIRS-based NF) training based on near-infrared spectroscopy would allow an improvement of the eating behavior, thus promoting a long-term weight loss in obese subjects.

Patients will be trained during a month with 8 NF sessions and results based on clinical data and different questionnaires results will be compared between inclusion and 3 months later

DETAILED DESCRIPTION:
Obesity is a disease of increasing prevalence due in part to the greater availability of fatty, sugary and/or salty foods which, when consumed chronically and in excess, can lead to food addiction.

According to the neurocognitive model of addiction, the development and maintenance of addiction is associated with deficits in cognitive control, as well as a decrease prefrontal cortex (dlPFC). Self-control in food choice situations also depends on prefrontal network with the dlPFC as a hub, strongly connected with striatal and cingulate structures.

Neurofeedback (NF) is a technique that relies on the patient's positive or negative self-regulation of brain activity. It has been shown to be effective in several pathologies, in particular attention deficit/hyperactivity disorder in young people and more recently in depression and emotion regulation.

In this study, NF will be based on near-infrared spectroscopy (fNIRS), because its use is easy mobile and inexpensive. The hypothesis is that the increase in dlPFC brain activity via fNIR-based NF training based on fNIRS would allow an improvement of the eating behavior, thus promoting a long-term weight loss in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for obesity surgery according to the 2009 French High Authority on Health (HAS) criteria (BMI ≥40 or BMI ≥35 with comorbidities)
* Right-handed
* Presenting a food addiction determined by the YFAS 2.0 questionnaire ;
* Affiliated to a social security system;
* Having given free and informed consent in writing.

Exclusion Criteria:

* Psychotic psychiatric disorders (schizophrenic disorders and bipolar disorders);
* Psychotropic drugs, except antidepressants stabilized for at least 3 weeks and benzodiazepines
* Addiction to alcohol or other psychoactive substances (except tobacco);
* History of bariatric surgery;
* Current treatment in the nutrition unit;
* Insufficient command of French;
* Pregnant or breast-feeding woman;
* Persons of legal age under legal protection (safeguard of justice, curatorship, guardianship), persons deprived of liberty.
* Contraindications to fMRI
* Inability to perform the fNIRS procedure due to blockage or attenuation of the light at the capillary level

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients who have a difference in resting state IRM after NF session | 1 month
  Difference in resting state IRM at inclusion and at 1 month after the 8th NF session between sham and experimental.
  Resting state IRM will allow to determine the correlation coefficient of the IRM BOLD signal fluctuations between the dlPFC and the striatum. The evolution of cognitive control by NeuroFeedback (NF) will thus be determined by a variation of this correlation coefficient and thus of the cortico-striatal connectivity at inclusion and after the 8th NF session.

SECONDARY OUTCOMES:
Number of patients who have a difference in resting state IRM after NF training in the cognitive food anticipation task condition | 1 month
  Variation in hemodynamic BOLD response in the cognitive food anticipation task condition between V1 and V8 between groups (NF vs sham).
  Difference in resting state IRM at inclusion and at 1 month after the 8th NF session between sham and experimental.
  Resting state IRM will allow to determine the correlation coefficient of the IRM BOLD signal fluctuations between the dlPFC and the striatum. The evolution of cognitive control by NeuroFeedback (NF) will thus be determined by a variation of this correlation coefficient and thus of the cortico-striatal connectivity at inclusion and after the 8th NF session.
Difference in blood pressure status 3 months after NF training | 4 months
  Evolution of health status using blood pressure (mmHg) between groups (NF vs sham) before and after participation (between V0 and V9).
Difference in blood pressure status 3 months after NF training | 4 months
  Evolution of health status using clinical exam criteria between groups (NF vs sham) before and after participation (between V0 and V9).
Difference in biological check up 3 months after NF training | 4 months
  Evolution of health status using biological check up between groups (NF vs sham) before and after participation (between V0 and V9).
Change of degree of correlation between EGG results and resting state IRM after NF training | 1 month
  Variation in the degree of correlation between electrogastrogramm plots and resting state MRI between V1 and V8 and between groups (NF vs sham).
Difference in mental Heath status after NF training between groups | 1 month
  Difference in anxiety and depression questionnaire (Hospital Anxiety and Depression Scale, questionnaire with 2 subscores, one for anxiety and one for depression. 0 = no anxiety/depression, 11 and more : anxiety/depression) after NF training between groups
Difference in mental Heath status training between groups after 3 months | 4 months
  Difference in anxiety and depression questionnaire (Hospital Anxiety and Depression Scale, questionnaire with 2 subscores, one for anxiety and one for depression. 0 = no anxiety/depression, 11 and more : anxiety/depression) 3 months after NF training between groups
Difference in Food frequency questionnaire scores between groups after NF training | 1 month
  Variation in FF questionnaire scores as a function of NF effect from inclusion to end of intervention.
  Food frequency questionnaire (FFQ) is a dietary assessment tool delivered as a questionnaire to estimate frequency and, in some cases, portion size information about food and beverage consumption over a specified period of time
Difference in Food Cravings Questionnaire-Trait-reduced scores between groups after NF training | 1 month
  Variation in Food Cravings Questionnaire-Trait-reduced scores as a function of NF effect from inclusion to end of intervention.
  Food Cravings Questionnaire (FCQ), which consists of a trait (FCQ-T; 39 items) and state (FCQ-S; 15 items) version. FCQ-T-r is a self-administrated questionnaire consisted of 15-items scored using a Likert-type scale (1 = never, 2 = rarely, 3 = sometimes, 4 = usually, 6 = always), for possible total scores ranging from 15 to 90.
Difference in Food Cravings Questionnaire-Trait-reduced scores between groups 3 months after NF training | 4 months
  Variation in Food Cravings Questionnaire-Trait-reduced scores as a function of NF effect from inclusion to 3 months after the end of intervention.
  Food Cravings Questionnaire (FCQ), which consists of a trait (FCQ-T; 39 items) and state (FCQ-S; 15 items) version. FCQ-T-r is a self-administrated questionnaire consisted of 15-items scored using a Likert-type scale (1 = never, 2 = rarely, 3 = sometimes, 4 = usually, 6 = always), for possible total scores ranging from 15 to 90.
Difference in Food frequency questionnaire scores between groups 3 months after NF training | 4 months
  Variation in Food Frequency questionnaire scores as a function of NF effect from inclusion to end of intervention.
  Food frequency questionnaire (FFQ) is a dietary assessment tool delivered as a questionnaire to estimate frequency and, in some cases, portion size information about food and beverage consumption over a specified period of time
Difference in Three Factor Eating Questionnaire-R18 scores between groups 3 months after NF training | 4 months
  Variation in Three Factor Eating Questionnaire-R18 questionnaire scores as a function of NF effect from inclusion to 3months after the end of intervention.
  The Three Factor Eating Questionnaire-R18 (TFEQ-R18) consists of 18 items on a 4-point response scale (definitely true/mostly true/mostly false/definitely false). Responses to each of the 18 items are given a score between 1 and 4 and item scores are summated into scale scores for cognitive restraint, uncontrolled eating, and emotional eating. Higher scores in the respective scales are indicative of greater cognitive restraint, uncontrolled, or emotional eating.
Difference in Three Factor Eating Questionnaire-R18 scores between groups after NF training | 1 month
  Variation in Three Factor Eating Questionnaire-R18 questionnaire scores as a function of NF effect from inclusion to the end of intervention.
  The Three Factor Eating Questionnaire-R18 (TFEQ-R18) consists of 18 items on a 4-point response scale (definitely true/mostly true/mostly false/definitely false). Responses to each of the 18 items are given a score between 1 and 4 and item scores are summated into scale scores for cognitive restraint, uncontrolled eating, and emotional eating. Higher scores in the respective scales are indicative of greater cognitive restraint, uncontrolled, or emotional eating.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rennes, Rennes, France